CLINICAL TRIAL: NCT01186107
Title: Randomized Comparison of Zotarolimus-Eluting Stent Versus Sirolimus-Eluting Stent Implantation for De Novo Coronary Artery DisEase in Patients With DIABETES Mellitus
Brief Title: Comparison of Zotarolimus-Eluting Stent vs Sirolimus-Eluting Stent for Diabetic Patients
Acronym: ESSENCE-DM2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D., Ph.D.,Professor of Medicine Asan Medical Center, University of Ulsan, College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-0220
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Disease; Diabetes
Keywords: coronary disease; stent
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endeavor Resolute stent (Experimental): zotarolimus-eluting stent
  Interventions: Device: Endeavor Resolute stent
- Cypher stent (Active Comparator): sirolimus-eluting stent
  Interventions: Device: Cypher stent

INTERVENTIONS:
Device: Endeavor Resolute stent — zotarolimus-eluting stent
  Arms: Endeavor Resolute stent
Device: Cypher stent — sirolimus-eluting stent
  Arms: Cypher stent

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of coronary stenting with the Zotarolimus-Eluting stent compared to the Sirolimus-Eluting stent in the treatment of de novo coronary stenosis in patients with diabetic patients.

DETAILED DESCRIPTION:
Prospective, two arms, single blind, randomized multi-center trial of 380 patients enrolled at 24 centers in Korea. Following angiography, diabetic patients with significant diameter stenosis >50% by visual estimation have documented myocardial ischemia or symptoms of angina, and eligible for stenting without any exclusion criteria will be randomized 1:1 to: a) Endeavor Resolute stent vs. b) Cypher select. All patients will be followed for at least 1 year. Angiographic follow-up at 9-months is routinely recommended.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with angina and documented ischemia
* Patients who are eligible for intracoronary stenting
* De novo lesion
* Percent diameter stenosis ≥50%
* Reference vessel size ≥ 2.5 mm by visual estimation

Exclusion Criteria:

* History of bleeding diathesis or coagulopathy
* Pregnant state
* Known hypersensitivity or contra-indication to contrast agent and heparin
* Limited life-expectancy (less than 1 year)
* Acute ST elevation myocardial infarction on admission
* Characteristics of lesion Left main disease In-stent restenosis Graft vessels
* Hematological disease (Neutropenia <3000/mm3, Thrombocytopenia <100,000/mm3)
* Hepatic dysfunction, liver enzyme (ALT and AST) elevation ≥ 3 times normal
* Renal dysfunction, creatinine ≥ 2.0mg/dL
* Contraindication to aspirin, clopidogrel or cilostazol
* Left ventricular ejection fraction <30%
* Patients who are actively participating in another drug or device - investigational study, which have not completed the primary endpoint follow- up period.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Angiographic in-segment late loss | 9-month angiographic follow-up

SECONDARY OUTCOMES:
Death (all-cause and cardiac) | at 12 months
myocardial infarction | at 12 months
stent thrombosis | at 12 months
target-lesion revascularization | at 12 months
target-vessel revascularization | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, Principal Investigator — Asan Medical Center
Locations (11):
- South Korea (11):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Kangwon University Hospital, Chuncheon
  - Daejeon St Mary's Hospital Catholic University, Daejeon
  - GangNeung Asan Hospital, Gangneung
  - Chonbuk National University Hospital, Jeonju
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Seoul Veterans Hospital, Seoul
  - Ulsan University Hospital, Ulsan